CLINICAL TRIAL: NCT05553730
Title: The Effects of Digital Buddy Programme on Older Adults' Mental Well-being: Study Protocol for a Multi-centre, Cluster Randomized Controlled Trial
Brief Title: Digital Buddy : Digital Inclusion for the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sally CHAN (Other)
Responsible Party: Sponsor-Investigator, Sally CHAN, President, Tung Wah College
Organization: Tung Wah College (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHI_0028_002
Record Dates: First submitted 2022-09-13; First posted 2022-09-23 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Mental Wellbeing of Older Adults

STUDY DESIGN:
Intervention Model Description: multi-centre, cluster randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Older adults randomly sorted into intervention group will receive six months of intervention after registration.
  Interventions: Behavioral: Digital Buddy program
- Control Group (No Intervention): Older adults randomly sorted into Control group will not receive six months of intervention after registration.

INTERVENTIONS:
Behavioral: Digital Buddy program — Six months of ICT and psychoeducation delivered by youth mentors via an e-learning platform
  Arms: Intervention Group

SUMMARY:
Digital exclusion is prominent in the older adult population in Hong Kong. Symptoms of depression and anxiety are shown to be linked with increased barriers to participate in society. It is essential for older adults to be digitally included, get prepared for the future challenges, make use of the online services offered by the Government and social organisations, and stay connected with families, friends and the wider world. The purposes of this study are to:

1. evaluate the effectiveness of a Digital Buddy program (digital literacy and psychoeducation training and interact with a young buddy for six-month period) on older adults' mental wellbeing, depressive symptoms, quality of life, self-efficacy and perceived social support; and
2. explore the perceptions of older adults and young buddie' perception of the Digital Buddy programme.

With one-to-one support from the young buddies, the older adults will be regularly using their digital device to communicate with family and friends, access to services available online, access to mental health and other healthcare information, more adherence to medication intake and easier to manage their health through health management/monitoring apps, and attend online activities organised by social organisations. It is hoped that by participating in this study, their mental well-being, self-efficacy and quality of life will be further improved. A long-term relationship is expected to build up among the young buddies and the older adults so that there would be ongoing social support for the older adults. Upon completion of this study, the toolkit will be made available to the public which can benefit the wider community.

DETAILED DESCRIPTION:
Study design:

This study will employ a multi-centre, cluster-randomized, two-parallel-group, controlled trial design with a 1:1 allocation ratio and no stratification. A total of 292 older adult participants and 30 young buddies will be recruited. Eligible older adults will be randomly assigned to intervention and control group. Intervention group will receive six months (a minimum of 23 hours) of digital literacy and psychoeducation training with a young buddy for six-month period. Under the guidance of a young buddy, older adult participants will learn and practice skills demonstrated in the video training courses and become familiarize with online health resources.

Intervention:

The Digital Buddy Program partners youth students from higher education institutions with older adults over the course of a six-month training program to help participants develop basic ICT skill and mental health knowledge. A new e-learning program will be developed which consists of video training courses, daily mood assessments and online health resources related to mental health and age-related conditions. The Program is expected to help older adults build confidence with navigating the internet and become familiarize with e-government resources and common social media platform, overcoming the barriers that prevent them from fully participating in society.

Study setting:

The study will be conducted in facilities for older people, including community centres and/or long-term care facilities for older adults in Hong Kong. Community centres for older adults provide various activities aiming to enable older adults to remain in the community and to lead a healthy, respectful and dignified life. Long-term care facilities for older adults provide residential care, meals, personal care, and nursing care for older adults who suffer from poor health or physical/mild mental disability.

Samples:

Convenience sampling approach will be used.

Intervention group:

The goal of the intervention is to enhance the ICT skills and promote the mental well-being of the older participants. A series of training sessions for a minimum of 23 hours will be provided to the older adults. In the training sessions, the Digital Buddy provides the older adults with educational support on some basic information and communication technology (ICT) skills and psychoeducation on some topics of mental health promotion.

The intervention will match up the older adults with the young adults (i.e., the Digital Buddy) in a ratio of 1 (young adults) to 10 (older adults). The study will recruit Digital Buddy if they are aged between 18 and 29 years and studying a full-time programme in a tertiary institution. The Digital Buddy will provide the training in flexible group size, at a flexible place, and at a flexible time aiming to accommodate the availability of both older and young adults. A train-the-trainer programme will be provided by the research team to the young adult participants. The young adult participants will be qualified to become Digital Buddies in this programme after they have completed the train-the-trainer programme. The contents of the train-the-trainer provide cover both the ICT skills and mental health promotion knowledge, as well as the essential communication skills with older people.

The training materials are uploaded to a newly developed web-based platform (www.twcdigitalbuddy.com.hk). This web-based platform contains all the educational materials related to ICT skills and mental promotion in various forms (e.g., video-based mini-lectures, micro-movies, and video-guided demonstrations). The educational materials are either newly produced by the team or already available on the web, yet they are all reviewed and content-validated by an expert panel. After equipping the older participants with the ICT skills so that they can independently exercise these skills to communicate with the Digital Buddy, the Digital Buddy will deliver the training sessions or necessary coaching on the e-platform (e.g., WhatsApp, Zoom). Both the older participants and the Digital Buddy will access the web-based training materials, attend the coaching, and communicate using smartphones.

To ensure satisfactory adherence to the intervention, the project team will telephone-contact both the Digital Buddy and the older participants at least once weekly to identify their difficulties participating in the intervention and solve their problems. To ensure the availability of access to the internet, older participants who do not own a smartphone will be provided with a smartphone with a data package complementarily during the study period.

Control group:

Participants in the group will receive the usual care. The research team will not provide any form of support to the participants in this group.

Participant timeline:

Participant recruitment and consenting will take place in the 4-week period before the baseline. Data collection of demographic and outcome data will take place at the baseline (T0). Interventions including the Digital Buddy and usual care will take place in the intervention period in week 1-24. Outcome data will be collected at week 25. Participants allocated to the usual care group will be given a waitlist intervention in week 26-49.

Recruitment:

Promotional seminars and booths will be conducted in the facilities for older adults (e.g., community centres for older people, residential care homes for older adults) and tertiary institutions. In the seminars, participants will be directly recruited. The programme will be introduced to collaborative organizations. Both printed and electronic posters will be produced and sent to the members of the collaborative organizations. The staff members of the collaborative organizations will help recruit their members to participate in this project.

Assignment of intervention:

Older participants after the completion of the eligibility assessment will be recruited. Data collection will be completed at baseline (T0). Participants completed the data baseline data collection will be randomly allocated to either the intervention or control groups in a 1:1 ratio. In the week after the completion of the intervention (T1), data collection on outcome markers will be implemented. Data of all participants in both groups will be employed for data analysis.

Cluster randomization method was employed to reduce the risk of within-cluster contamination because most of the training materials are open source that participants are share within their peers in a cluster. A permuted block (block size=4) random allocation sequence list with an allocation ratio to either intervention group or control at 1:1 will be generated by the web-based application www.random.org. The cluster unit of randomization is based on a facility for older adults (e.g., one community centre as a unit). Each unit will be randomly assigned after the entire unit is screened, written consent is obtained, and baseline assessment is completed to reduce the risk of selection bias. A group of four units (i.e., the size of a permuted block) with a similar number of eligible and consented participants will be grouped to be randomly allocated. This aims to ensure each group comprises a similar number of participants. The random allocation process will be implemented by an independent statistician, who will not participate in any other parts of the proposed study. The statistician will assign group labels to each unit based on their sequence of entries with reference to the sequence list, thus ensuring that other members of the research team cannot foresee the group allocations. In this study, only the outcome assessor will be blinded to the group labels. It will not be possible to blind the participants or the interventionists.

A waitlist control design will be adopted so that the participants randomized into the control group will be provided with a chance to receive the intervention after they have completed their untreated condition (i.e., receiving usual care for six months).

Oversight and monitoring:

A trial steering team of three academics in the disciplines of nursing and occupational therapy will direct the whole study process. The project implementation team comprising one project officer and one project assistant will be responsible to provide day-to-day support for the trial. An advisory panel comprising one geriatrician and one social worker specialising in gerontology will provide advice to the project. The trial steering team will meet the project implementation team bi-week to monitor the quality of implementation. The advisory panel will meet the trial steering team once per three months to advise on upholding the quality of the trial.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years or above,
* able to speak Cantonese and read Chinese,
* mentally capacitated is defined as having no diagnosed mental diseases leading to being mentally disabled and certified by a psychiatrist

Exclusion Criteria:

* unable to communicate in Cantonese.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Five Well Being Index (WHO-5) at 6 months | Collected at T0 (baseline) and T1 (i.e., the week six months after the completion of the intervention
  The World Health Organization Five Well-being Index (WHO-5) will be used to measure mental well-being over the past two weeks. WHO-5 comprises five items and each item is rated by a 6-point Likert scale from 0 (at no time) to 5 (all of the time). The total score ranges from 0 to 25. A higher score indicates an increased sense of psychological well-being. The Cantonese version of WHO-5 showed good internal consistency (α=0.86) and good concurrent validity with quality of life (r=0.41-0.51).
Change from Baseline 9-item Patient Health Questionnaire - 9 (PHQ-9) at 6months | Collected at T0 (baseline) and T1 (i.e., the week six months after the completion of the intervention
  The 9-item Patient Health Questionnaire (PHQ-9) will be used to measure depressive symptoms over the past two weeks. PHQ-9 comprises nine items and each item is rated by a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 27. A higher score indicates greater severity of depressive symptoms. The Cantonese version of PHQ-9 showed good internal consistency (α=0.82), test-retest reliability (r=0.76), and satisfactory concurrent validity with the mental component of quality of life (r=-0.60).
Change from Baseline 12-item Short Form survey version 2 (SF-12v2) at 6 months | Collected at T0 (baseline) and T1 (i.e., the week six months after the completion of the intervention
  The version 2 of the 12-item Short Form Health Survey (SF-12v2) will be used to measure health-related quality of life over the past four weeks. SF-12v2 comprises 12 items rated by scales with varying points measuring eight domains of health, including physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The scores of eight domains are aggregated into two scores: 1) physical component summary score and 2) mental component summary score. The scores will be calculated by a standard algorithm. A higher component summary scores indicates a better health-related quality of life. The Chinese version of SF-12v2 showed good test-retest reliability (r=0.67-0.82), good construct validity with >80% of total variance explained by the two-factor model.
Change from Baseline 10-item General Self-Efficacy Scale (GSES-10) at 6 months | Collected at T0 (baseline) and T1 (i.e., the week six months after the completion of the intervention
  The 10-item General Self-efficacy scale (GSES-10) will be used to measure self-efficacy. GSES-10 comprises 10 items and each item is rated by a 4-point Likert scale from 1 (not at all true) to 4 (exactly true). The total score ranges from 10 to 40. A higher score indicates better self-efficacy. The Chinese version GSES-10 showed good internal consistency (α=0.91), good criterion validity with wellbeing (r=0.56-0.63, p<0.001), self-esteem (r=0.40-0.49, p<0.001), and mental health (0.39-0.41, p<0.001).
Change from Baseline Multidimensional Scale of Perceived Social Support (MSPSSC) at 6 months | Collected at T0 (baseline) and T1 (i.e., the week six months after the completion of the intervention
  The 12-item Multidimensional Scale of Perceived Social Support (MSPSS) will be used to measure perceived social support. MSPS comprises 12 items which are factored in three subscales by sources of support (i.e., family, friends, significant others). Each subscale comprises four items. Each item is rated on a 7-point Likert scale from 1 (strongly disagree) to 7 (strongly agree). The total score ranges from 12 to 84. A higher score indicates better social support. The Chinese version of MSPSS showed good internal consistency (Cronbach's α=0.95), good test-retest reliability (ICC=0.91), and satisfactory concurrent validity with perceived stress (r=-0.221) and caregiving rewarding feelings (r=-0.327).

CONTACTS AND LOCATIONS:
Overall Officials: Sally Chan, Principal Investigator — Tung Wah College
Locations (1):
- Tung Wah College, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Kwan RYC, Ng F, Lai M, Tsien-Wong TBK, Leung EMF, Chan S. The effects of the Digital Buddy programme on mental health in older adults: A multi-centre, cluster randomised controlled trial. Digit Health. 2026 Feb 6;12:20552076261419978. doi: 10.1177/20552076261419978. eCollection 2026 Jan-Dec. PMID 41659058
- [Derived] Kwan RYC, Ng F, Lai M, Wong D, Chan S. The effects of Digital Buddy programme on older adults' mental well-being: study protocol for a multi-centre, cluster randomized controlled trial. Trials. 2023 Feb 7;24(1):95. doi: 10.1186/s13063-023-07130-5. PMID 36750879